CLINICAL TRIAL: NCT05081466
Title: Associations Between Diet and Hip Fracture Incidence in the United Kingdom Women's Cohort
Brief Title: Diet and Hip Fracture Risk in the United Kingdom Women's Cohort
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Darren Greenwood, Senior Lecturer in Biostatistics, University of Leeds
Other Study IDs: HRA 17/YH/0144
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Hip Fracture (First Incidence of)
Keywords: Nutrition; Fracture; Cohort study; Epidemiology; Osteoporosis
MeSH Terms: conditions — Hip Fractures; Fractures, Bone; Osteoporosis | interventions — Dietary Patterns; Fruit; Tea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- United Kingdom Women's Cohort: United Kingdom Women's Cohort Study. No interventions are to be administered in this observational prospective cohort study.
  Interventions: Other: Dietary pattern; Other: Fruit and vegetable intake; Other: Meat intake; Other: Fish intake; Other: Egg intake; Other: Dairy intake; Other: Tea intake; Other: Coffee intake; Other: Tea and coffee intake; Other: Protein intake; Other: Calcium intake; Other: Vitamin D intake

INTERVENTIONS:
Other: Dietary pattern — (regular meat-eater, occasional meat-eater, fish-eater, vegetarian, and vegan)
Other: Fruit and vegetable intake — Intake of fruits, vegetables, fruits and vegetables combined from food frequency questionnaire
Other: Meat intake — Red meat, poultry, processed meat from food frequency questionnaire
Other: Fish intake — Intake of fish from food frequency questionnaire
Other: Egg intake — Intake of eggs from food frequency questionnaire
Other: Dairy intake — Intake of dairy products from food frequency questionnaire
Other: Tea intake — Intake of tea (drink) from food frequency questionnaire
Other: Coffee intake — Intake of coffee (caffeinated or decaffeinated) from food frequency questionnaire
Other: Tea and coffee intake — Combined intake of tea and coffee from food frequency questionnaire
Other: Protein intake — Estimated intake of protein, derived from food frequency questionnaire
Other: Calcium intake — Estimated intake of calcium, derived from food frequency questionnaire
Other: Vitamin D intake — Estimated intake of vitamin D, derived from food frequency questionnaire and any recorded supplemental intake

SUMMARY:
Hip fracture is a common serious injury in older women that reduces quality of life and can lead to premature death. In the United Kingdom, hip fractures are estimated to account for 1.5 million hospital bed days used per year due to long hospitalisation and rehabilitation periods post-surgery, costing the National Health Service over £1 billion per year. Diet can affect bone health and risk of hip fracture, with varying risks in women on specific diets, and specific foods and nutrients playing more important roles than others. Vegetarians may be at a greater risk of hip fracture than meat-eaters, and those who don't consume enough protein could be at a greater risk than those with adequate intakes. This research aims to investigate which dietary factors (and in what quantities) might predispose United Kingdom women to a greater risk of hip fracture, and which factors may be protective. The purpose of this study is to better understand the role of diet in reducing hip fracture risk in United Kingdom women. The research will use existing dietary and lifestyle data from the United Kingdom Women's Cohort Study and hospital records of hip fractures.

DETAILED DESCRIPTION:
Background: Hip fracture is an increasingly prevalent global health condition that increases morbidity and mortality. Previous observational studies have shown potential for risk reduction through diet modification, but associations between many dietary factors and hip fracture incidence are uncertain, and evidence in United Kingdom populations is limited. Therefore, this study aims to assess associations between diet and hip fracture incidence in the United Kingdom Women's Cohort.

Research plan and methods: The investigators will utilise dietary and lifestyle data from the United Kingdom Women's Cohort which recruited 35,372 middle-aged women between 1995-1998. This data has been linked with Hospital Episode Statistics to provide hip fracture data of participants.

Cox regression models will be applied to explore potential associations between dietary factors and hip fracture incidence. Dietary factors will be modelled both as categorical and continuous so that models can be fit comparing the risk of hip fracture between categories of intakes and per increment increase in exposure intake (linear dose-response). Cubic splines will be used to model non-linear associations for dietary intake of fruits, vegetables, tea, and coffee since previous research has suggested possible non-linear associations for these variables.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 35 - 69 years at time of recruitment
* Able to provide informed consent

Exclusion Criteria:

* Male
* Not a resident of England
* Unable to link dietary and lifestyle data with hospital episode data
* Missing covariate data
* Hip fracture or osteoporosis prevalence before or on the date of recruitment

Ages: 36 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The UK Women's cohort profile is published here: [https://doi.org/10.1093/ije/dyv173].
Sampling Method: Probability Sample
Enrollment: 35372 (Actual)
Dates: Start 1995-01-15 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Hip fracture incidence (first) | age when the completed questionnaire was returned (1995-1998) until age at event, death, or end of study period (19 Mar 2019)
  Incidence of first hip fracture ascertained from linkage to Hospital Episode Statistics (HES) data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Webster J, Greenwood DC, Cade JE. Risk of hip fracture in meat-eaters, pescatarians, and vegetarians: results from the UK Women's Cohort Study. BMC Med. 2022 Aug 11;20(1):275. doi: 10.1186/s12916-022-02468-0. PMID 35948956
- [Derived] Webster J, Greenwood DC, Cade JE. Foods, nutrients and hip fracture risk: A prospective study of middle-aged women. Clin Nutr. 2022 Dec;41(12):2825-2832. doi: 10.1016/j.clnu.2022.11.008. Epub 2022 Nov 9. PMID 36402009

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT05081466/SAP_000.pdf